CLINICAL TRIAL: NCT01105546
Title: An Investigator-initiated Study on rFVIIa Prophylaxis in Children With Hemophilia A and Inhibitors - European Initiative to Prevent Joint Damage in Hemophilia A Children With Inhibitors
Brief Title: rFVIIa Prophylaxis in Children With Hemophilia A and Inhibitors
Acronym: ENJOIH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Elena Santagostino, MD, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENJOIH 01; IND 14503 (Other: FDA)
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Hemophilia A With Inhibitors
Keywords: hemophilia A; inhibitors; prophylaxis; immune tolerance induction
MeSH Terms: conditions — Hemophilia A | interventions — recombinant FVIIa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prophylaxis (Experimental): prophylaxis with recombinant activated FVII 90 µg/kg/day i.v.
  Interventions: Drug: recombinant activated factor VII
- on demand treatment (Active Comparator): treatment of bleeding episodes with 270 µg/kg (first/single dose) or 90 µg/kg i.v. every 2-3 hours until bleeding resolution
  Interventions: Drug: recombinant activated factor VII

INTERVENTIONS:
Drug: recombinant activated factor VII — 90 µg/kg/day i.v.
  Other Names: NovoSeven
  Arms: prophylaxis
Drug: recombinant activated factor VII — treatment of bleeding episodes with 270 µg/kg (first/single dose) or 90 µg/kg i.v. every 2-3 hours until bleeding resolution
  Other Names: NovoSeven
  Arms: on demand treatment

SUMMARY:
The study evaluates the efficacy and safety of a prophylactic treatment with recombinant activated FVII in reducing the frequency of joint bleeds and the development of joint damage in children with hemophilia A who develop high-titer inhibitors.

DETAILED DESCRIPTION:
This is a multicentre, randomised, controlled study designed to gain evidence of the advantage of the prophylactic, daily treatment with recombinant activated FVII as compared to the conventional on demand therapy in reducing the bleeding frequency and preserving the orthopaedic status in hemophilic children with inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemophilia A who have been treated with factor VIII on demand or on prophylaxis and who have developed inhibitors to factor VIII
* ≤ 2 years from the time of first inhibitor detection.
* High-responding inhibitors (historical peak > 5 BU/mL)and known anamnestic response in case of negative inhibitor titre.
* Candidates to start daily ITI with FVIII doses ranging from 50 IU/Kg/day to 200 IU/Kg/day
* Maximal two bleedings in the same joint within the last 6 months before entering the study or maximal six joint bleeds in the same joint within 2 years
* Adequate venous access for daily infusion and capable (caregiver) of reconstituting and injecting the study drug
* Informed consent by parents or legal guardians.

Exclusion Criteria:

* ITI already started
* Known or suspected hypersensitivity to the active substance or to any of the excipients of the study drug
* Administration of any investigational product within 30 days prior to randomisation
* Other coagulation disorders than congenital hemophilia A.
* Family history of thrombosis at an early age (< 40 years), known thrombophilia, any previous thrombosis including catheter-related deep vein thrombosis, previous neonatal thrombosis.
* Known pseudo tumours
* Known severe liver disease
* Platelet count < 50,000 platelets/µL at screening
* Surgery within one month or planned major and/or orthopaedic surgery.

Max Age: 8 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-02 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Total number of joint bleeds. | 18 months

SECONDARY OUTCOMES:
Joint status evaluated by the Hemophilia Joint Health Score | 18 months
Number of adverse events and serious adverse events. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Elena Santagostino, MD, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (15):
- United States (3):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Children's Mercy Hospital, Kansas City, Missouri
- Haemophilia Comprehensive Care Centre, Edouard Herriot University Hospital, Lyon, France
- Germany (3):
  - Vivantes Klinikum im Friedrichshain Haemophilia Care Center, Medical Center, Berlin, Germany
  - Klinikum Bremen-Mitte, Prof.-Hess-Kinderklinik, Bremen
  - Klinikum der Johann Wolfgang Goethe-Universitat, Frankfurt/M
- Italy (3):
  - Angelo Bianchi Bonomi Hemophilia and Thrombosis Center, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy
  - Azienda Ospedaliero-Universitaria Careggi Agenzia per l'emofilia e Centro di riferimento regionale per i disordini congeniti del sanguinamento, Florence
  - Centro Emofilia e Trombosi Unità Operativa di Ematologia Ospedale San Giovanni Bosco, Napoli
- Romania (2):
  - National Institute for Transfusional Hematology, Bucharest, Romania
  - Spitaluc Clinic de Urgenta pentru Copii Louis Turcanu, University of Medicine and Pharmacy, Timișoara, Romania
- Spain (3):
  - Unitat Hemofilia, Hospital Vall d'Hebron, Barcelona, Spain
  - Centro de Hemofilia, Hospital Universitario La Paz, Madrid, Spain
  - Unidad de Coagulopatias Congenitas, Hospital Universitario la Fe, Valencia, Spain